CLINICAL TRIAL: NCT05032924
Title: The Clinical and Biological Effect of Extracorporeal Shock Wave Technology (ESWT) With Combined PRP Therapy on Rotator Cuff Lesions
Brief Title: The Clinical and Biological Effect of ESWT With Combined PRP Therapy on Rotator Cuff Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Jih-Yang Ko, Professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202100718A3A3
Record Dates: First submitted 2021-08-03; First posted 2021-09-02 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Rotator Cuff Lesions
Keywords: Platelet Rich Plasma (PRP); Extracorporeal shock wave therapy (ESWT)

STUDY DESIGN:
Intervention Model Description: Participants are randomly into four group to receive either shockwave or PRP or sham (HA) treatment based on a computerized statistical randomization. Every participant will have Subacromial injection of 2.5 ml PRP form Regen Kit BCT 1 or HA (control)(HYAJOINT Synovial Fluid Supplement, active ingredient: Sodium Hyaluronate 25 mg, package: 2.5 mL per syringe) one week before ESWT or sham therapy.
  Follow-up examinations are performed independently by one of the coauthors, who is blinded to patient treatment status at 1week, 2week, 1month, 3 months, 6 months, and 12 months after treatment. Peripheral blood (10cc) will be collected one week and 1 month after treatment and shoulder MRI will be checked 12 months after treatment. Participants who have persistent shoulder discomfort may be advised to undergo surgical intervention.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PPR group (Experimental): Receive PRP injection only (PRP form Regen Kit BCT 1)
  Interventions: Combination Product: PPR group with ESWT; Combination Product: PPR group without ESWT
- HA group (Placebo Comparator): Receive HA injection only (HYAJOINT Synovial Fluid Supplement, active ingredient: Sodium Hyaluronate 25 mg, package: 2.5 mL per syringe)
  Interventions: Combination Product: HA group with ESWT; Combination Product: HA group without ESWT

INTERVENTIONS:
Combination Product: PPR group with ESWT — extracorporeal shock wave (ESWT) (STORZ MEDICAL Extracorporeal Shock Wave Therapy) (3000 impulse, each point, 24 KV, 0.32 mJ/mm2) one week after PRP or HA injection
  Arms: PPR group
Combination Product: PPR group without ESWT — PRP or HA injection only
  Arms: PPR group
Combination Product: HA group with ESWT — extracorporeal shock wave (ESWT) (STORZ MEDICAL Extracorporeal Shock Wave Therapy)
  Arms: HA group
Combination Product: HA group without ESWT — PRP or HA injection only
  Arms: HA group

SUMMARY:
Through the investigators previous study of the effect of transient increased cellular permeability after ESWT, combined ESWT and PRP may have better effect on the treatment of rotator cuff lesions. The investigators intend to conduct a prospective double blind randomized control study on the treatment effect of combined ESWT and PRP therapy for rotator cuff lesions without complete tearing. Constant Score, VAS and data from peripheral blood will be measured for the effectiveness evaluation. Shoulder MRI will be followed-up one year after ESWT. The investigators hypothesize that combined ESWT and PRP will be more effective for rotator cuff lesions.

DETAILED DESCRIPTION:
Overall Design [Prospective randomized double-blind study for the clinical effect of combined ESWT and platelet-rich plasma (PRP) or PRP or ESWT alone or sham treatment on patients with shoulder rotator cuff lesions and without complete tear.]

The participants will be separated into 4 groups according to computer statistical randomization.

The investigators shall use STORZ MEDICAL Extracorporeal Shock Wave Therapy 3000 impulse 24KV (0.32mJ/mm2) Focus at two points (3000 impulse each point) near the insertion of supraspinatus and rotation interval of the involved shoulder.

PRP： The PRP form Regen Kit BCT 1 Platelet Rich Plasma PRP will be used and will be injected into the Subacromial bursa (Hyajoint injection as a control)

HYAJOINT Synovial Fluid Supplement, active ingredient: Sodium Hyaluronate 25 mg, package: 2.5 mL per syringe

The randomized, double-blind, placebo-controlled clinical study will involve 30-50 patients who have rotator cuff lesions without complete tear. The inclusion criteria are (1) patients who have pain around the shoulder, a positive impingement sign, and a positive imaging diagnosis of rotator cuff pathology without complete tear; (2) patients who do not respond to conservative therapy or rehabilitation for at least 3 months; and (3) patients age between 35 and 80 years, who sign the informed consent form. The investigators will exclude patients who have rheumatic diseases, glenohumeral osteoarthritis, full-thickness cuff tears, fractures, infections, or tumors; those who have received a subacromial injection within 3 weeks; and those who are pregnant or want to become pregnant; and those who have arrhythmia, pacemaker, coagulopathy, or malignancy.

The intent-to-treat population is a fully randomized group of patients who have a baseline value (Constant score and VAS before treatment). The imaging diagnosis of a rotator cuff lesion is made by a musculoskeletal radiologist who has considerable experience in interpreting magnetic resonance imaging (MRI) results for shoulders. On MRI, rotator cuff tendinosis is characterized by increased in tratendinous signal intensity onT2-weighted images without tendon disruption. The tendinosis of the MRI imaging was further diverted into three grades. Grade 1 indicates less than 1/3 of the supraspinatus tendon is involved, Grade 2 indicates 1/3 to 2/3 and Grade 3 indicates more than 2/3 of the supraspinatus tendon is involved. Partial-thickness tearing is characterized by the presence of focal hyperintense fluid or a fluid-like signal intensity that extended into the tendon on the T2-weighted images. A full thickness tear is diagnosed by the extension of hyperintense fluid or fluid-like signal intensity through the entire thickness of the interrupted rotator cuff tendon on T2-weighted images.

Every participant will have Subacromial injection of 2.5 ml PRP or HA (control) one week before ESWT or sham therapy. In Group I, patients receive 3000 impulses of shockwaves at 24kV (energy flux density, 0.32mJ/mm2) to the affected shoulder as a 1-time treatment. Treatments are performed on an outpatient basis. The area of treatment (2 points near the supraspinatus insertion and rotator interval) is focused with a control guide on the machine, and surgical lubricant is placed on the skin in contact with the shockwave tube with the patient in a supine position. The sham treatment entail use of the device in which the silicone pad was removed from the stand-off device, but the participants can still hear the sound of the shock wave and have tingling sensation over the skin but without energy transduced. The participants' vital signs and local discomfort are monitored throughout the course of treatment. The treated area is inspected for local swelling, ecchymosis, or hematoma immediately after the treatment.

The participants will have a pain medication-free interval 3 days prior to each evaluation. After treatment and during follow-up, participants will be restricted to the use of a 750mg of acetaminophen per day for pain, in order to facilitate usage and comparison of the medications among the patients. Follow-up examinations are performed independently by one of the coauthors, who is blinded to patient treatment status at 1week, 2week, 1month, 3 months, 6 months, and 12 months after treatment. Peripheral blood (10cc) will be collected one week and 1 month after treatment and shoulder MRI will be checked 12 months after treatment. The participants who have persistent shoulder discomfort may be advised to undergo surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

1. pain around the shoulder, a positive impingement sign, imaging diagnosis of rotator cuff pathology without complete tear
2. do not respond to conservative therapy or rehabilitation for at least 3 months
3. age between 35 and 80 years, who sign the informed consent form.

Exclusion Criteria:

1. rheumatic diseases, SLE, diabetic neuropathy, glenohumeral osteoarthritis, full-thickness cuff tears, fractures, infections, or tumors
2. received a subacromial injection within 3 weeks
3. pregnant or want to become pregnant.
4. arrhythmia, pacemaker, coagulopathy, or malignancy

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-08-02 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Constant Score | measure and record at 1 month after treatment.
  The Constant Score contains pain (15 points), activities of daily living (20 points), mobility (40 points), and strength (25 points). Improve the Constant Score by 10 points for treatment success. For monitoring the participants' recovery progress, will measure and record at 1 month after treatment.
Constant Score | measure and record at 3 months after treatment.
  The Constant Score contains pain (15 points), activities of daily living (20 points), mobility (40 points), and strength (25 points). Improve the Constant Score by 10 points for treatment success. For monitoring the participants' recovery progress, will measure and record at 3 months after treatment.
Constant Score | measure and record at 6 months after treatment.
  The Constant Score contains pain (15 points), activities of daily living (20 points), mobility (40 points), and strength (25 points). Improve the Constant Score by 10 points for treatment success. For monitoring the participants' recovery progress, will measure and record at 6 months after treatment.
Constant Score | measure and record at 12 months after treatment.
  The Constant Score contains pain (15 points), activities of daily living (20 points), mobility (40 points), and strength (25 points). Improve the Constant Score by 10 points for treatment success. For monitoring the participants' recovery progress, will measure and record at 12 months after treatment.
visual analog scale (VAS) | measure and record at 1 month after treatment.
  Assess whether the pain level is reduced. The VAS with two endpoints representing 0 ('no pain') and 10 ('extreme pain'). For monitoring the patients' recovery progress, will measure and record at 1 month after treatment.
visual analog scale (VAS) | measure and record at 3 months after treatment.
  Assess whether the pain level is reduced. The VAS with two endpoints representing 0 ('no pain') and 10 ('extreme pain'). For monitoring the patients' recovery progress, will measure and record at 3 months after treatment.
visual analog scale (VAS) | measure and record at 6 months after treatment.
  Assess whether the pain level is reduced. The VAS with two endpoints representing 0 ('no pain') and 10 ('extreme pain'). For monitoring the patients' recovery progress, will measure and record at 6 months after treatment.
visual analog scale (VAS) | measure and record at 12 months after treatment.
  Assess whether the pain level is reduced. The VAS with two endpoints representing 0 ('no pain') and 10 ('extreme pain'). For monitoring the patients' recovery progress, will measure and record at 12 months after treatment.
Range of Motion (ROM) | measure and record at 1 month after treatment.
  Assess whether the range of motion is increased. Measure the motions: abduction, elevation through flexion, external rotation and internal rotation. For monitoring the patients' recovery progress, will measure and record at 1 month after treatment.
Range of Motion (ROM) | measure and record at 3 months after treatment.
  Assess whether the range of motion is increased. Measure the motions: abduction, elevation through flexion, external rotation and internal rotation. For monitoring the patients' recovery progress, will measure and record at 3 months after treatment.
Range of Motion (ROM) | measure and record at 6 months after treatment.
  Assess whether the range of motion is increased. Measure the motions: abduction, elevation through flexion, external rotation and internal rotation. For monitoring the patients' recovery progress, will measure and record at 6 months after treatment.
Range of Motion (ROM) | measure and record at 12 months after treatment.
  Assess whether the range of motion is increased. Measure the motions: abduction, elevation through flexion, external rotation and internal rotation. For monitoring the patients' recovery progress, will measure and record at 12 months after treatment.
MRI | shoulder MRI will be checked 12 months after treatment
  Take shoulder MRI to compare the difference before and after treatment. The degeneration of the supraspic is graded as: grade 1 ≤ 1/3; 1/3 < grade 2 < 2/3; grade 3 ≥ 2/3.

CONTACTS AND LOCATIONS:
Overall Officials: Jih-Yang Ko, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Medical Hosptial, Kaohsiung City, Taiwan